CLINICAL TRIAL: NCT00371137
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study of Xyrem® in Subjects With Fibromyalgia
Brief Title: A Safety and Efficacy Study of Xyrem® in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-008
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Fibromyalgia
Keywords: FMS; Fibro; pain; Body pain; tenderness; joint pain; stiffness; muscular pain
MeSH Terms: conditions — Fibromyalgia; Pain; Arthralgia; Myalgia | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Xyrem®

INTERVENTIONS:
Drug: Xyrem® — two doses
  Arms: 2
Drug: Placebo — Oral Solution
  Arms: 1

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of Xyrem® compared to placebo for the treatment of fibromyalgia in a randomized, double blind, placebo controlled, parallel group trial.

DETAILED DESCRIPTION:
The trial is a randomized, double blind, placebo controlled, parallel group trial in subjects diagnosed with fibromyalgia in accordance with the American College of Rheumatology. Total duration is up to twenty-one (21) weeks of trial participation. Subjects will undergo a screening and withdrawal/washout period lasting up to five (5) weeks combined, followed by baseline period lasting one (1) week. Total treatment duration will be fourteen (14) weeks followed by one (1) week safety follow-up post treatment period. During the screening and withdrawal/washout period, no study medication will be given; however rescue medication acetaminophen (up to 4 grams per day) will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years or older who meet the American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia.

Exclusion Criteria:

* Subjects will be excluded if they have a history of rheumatic disease or other disorders that may compromise reliable representation of subjective symptoms.
* Any other condition that will cause a risk to subjects if they participate in the trial is also a reason for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I. Jon Russell, PhD, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (70):
- United States (70):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Rheumatology Associates of N. AL, PC, Huntsville, Alabama
  - Xenoscience, Inc. dba 21st Century Neurology, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Providence Clinical Research, Burbank, California
  - Northern California Research, Carmichael, California
  - Pasadena Rehabilitation Institute, Pasadena, California
  - Arroyo Medical Group, Pismo Beach, California
  - Sacramento Research Medical Group, Sacramento, California
  - Apex Research Institute, Santa Ana, California
  - Sansum Clinic, Santa Barbara, California
  - Robert E. Harris, MD Medical Corporation, Whittier, California
  - CRIA Research, Fort Lauderdale, Florida
  - Clinical Physiology Associates Clinical Study Center, Fort Meyers, Florida
  - Innovative Research, Largo, Florida
  - Compass Research, Orlando, Florida
  - Sunrise Medical Research, Plantation, Florida
  - Coastal Medical Research, Inc, Port Orange, Florida
  - Deerpath Physicians Group, Gurnee, Illinois
  - Balanced health Research Center, Peoria, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Graves - Gilbert Clinic, Bowling Green, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Commonwealth Biomedical Reseach, LLC, Madisonville, Kentucky
  - FutureCare Studies, Springfield, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - PCM Medical Services, Lansing, Michigan
  - Clinvest, Springfield, Missouri
  - Clayton Medical Associates, St Louis, Missouri
  - St. John's Mercy Health System, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - CCR Trials, Berlin, New Jersey
  - School of Osteopathic Medicine, Cherry Hill, New Jersey
  - Anderson & Collins Clinical Research, Inc., Edison, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - AAIR Research Center, Rochester, New York
  - Great Lakes Medical Research, Westfield, New York
  - Carolina Bone and Joint, Charlotte, North Carolina
  - Carolinas Research, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Radiant Research, Columbus, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Radiant Research, Mogadore, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - PRO Research, Eugene, Oregon
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Low Country Research Center, Charleston, South Carolina
  - Radiant Research, Greer, Greer, South Carolina
  - Clinsearch, Chattanooga, Tennessee
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Walter M. Chase, MD, Austin, Texas
  - Future Search Trials of Neurology Future Research Trials, Austin, Texas
  - DFW Wellness, Fort Worth, Texas
  - The Methodist Hospital Systems, Houston, Texas
  - Houston Sleep Center, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - Fatigue Consultation Center, Salt Lake City, Utah
  - Richard A. Neiman, MD, Inc., Kirkland, Washington
  - Pacific Rheumatolgy Associates, Inc., Renton, Washington
  - Charrleston Internal Medicine, Charleston, West Virginia

REFERENCES:
- [Result] Russell JI, Holman AJ, Swick TJ, Alvarez-Horine S, Wang GY, Guinta D; Sodium Oxybate 06-008 FM Study Group. Sodium oxybate reduces pain, fatigue, and sleep disturbance and improves functionality in fibromyalgia: results from a 14-week, randomized, double-blind, placebo-controlled study. Pain. 2011 May;152(5):1007-1017. doi: 10.1016/j.pain.2010.12.022. Epub 2011 Mar 11. PMID 21397402
- [Result] Swick TJ, Alvarez-Horine S, Zheng Y, Rothman J, Inhaber N, Holman AJ, Smith TR, Russell IJ. Sodium Oxybate Improves Pain, Fatigue, and Sleep in Fibromyalgia: Results from a 14-Week Randomized, Double-Blind, Placebo-Controlled Trial. [APSS abstract 0984]. Sleep 2009;32(suppl):A321.
- [Result] Swick TJ, Alvarez-Horine S, Zheng Y, Guinta D, Inhaber N, Holman AJ, Smith TR, Russell IJ. Impaired Sleep and Daytime Functioning at Baseline in Subjects with Fibromyalgia from a 14-Week Randomized, Double-Blind, Placebo-Controlled Trial of Sodium Oxybate. [APSS abstract 1013]. Sleep 2009;32(suppl):A330.
- [Result] Mease PJ, Swick TJ, Alvarez-Horine S, Inhaber N, Guinta DR, Holman AJ, and Russell IJ. Sodium Oxybate Improves Fatigue, Sleep Disturbance, and PGIC in Fibromyalgia-Results form a Phase 3, 14-Week, Controlled Trial. Arthritis & Rheum 2009;60(10):S529.
- [Result] Russell IJ, Alvarez-Horine S, Zheng Y, Guinta DR, Holman AJ and Swick TJ. Effect of Sodium Oxybate on Pain, PGIC, & Composite Scores in Fibromyalgia-Results from a Phase 3 Controlled Trial. Arthritis & Rheum 2009;60(10):S528.
- [Result] Swick TJ, Rosenfeld V, Alvarez-Horine S, Guinta D, Wang YG, Russell IJ. Improvement in Multiple Symptoms of Fibromyalgia With Sodium Oxybate Treatment: Results From a US Phase 3 Randomized, Controlled Trial [AAN abstract P03.292]. Neurology. 2010;74(suppl 2):A279.
- [Result] Jones KD, Bennett RM, Alvarez-Horine S, Wang YG, Guinta D, Russell IJ. Sodium Oxybate Improves Function and Quality of Life in Fibromyalgia-Results From a Phase 3, Randomized, Controlled Trial [APS abstract 262]. J Pain. 2010;11(suppl 1):S41.
- [Result] Russell IJ, Perkins AT, Michalek JE; Oxybate SXB-26 Fibromyalgia Syndrome Study Group. Sodium oxybate relieves pain and improves function in fibromyalgia syndrome: a randomized, double-blind, placebo-controlled, multicenter clinical trial. Arthritis Rheum. 2009 Jan;60(1):299-309. doi: 10.1002/art.24142. PMID 19116896
- [Result] Silverman S, Holman AJ, Benson B, Alvarez-Horine S, Wang YG, Sarzi-Puttini. Sodium Oxybate Improves Sleep and Fatigue in Patients With Fibromyalgia: Pooled Analysis From 2 Pivotal Clinical Trials [ACR/ARHP abstract 2337]. Arthritis Rheum. 2010;62(suppl 10):815.
- [Result] Spaeth M, Russell IJ, Perrot S, Choy E, Benson B, Wang YG, Lai C. The Effects of Sodium Oxybate on Multiple Symptoms of Fibromyalgia: Results From Two Phase 3, Randomized, Double-Blind, Controlled Trials. In: Myopain 2010 Abstracts; October 3-7, 2010; Toledo, Spain. Abstract 39.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo taken as two equally divided nightly doses
- Xyrem 4.5g: Xyrem 4.5g taken as two equally divided nightly doses
- Xyrem 6.0g: Xyrem 6.0g taken as two equally divided nightly doses
Period: Overall Study
Arm/Group | Placebo | Xyrem 4.5g | Xyrem 6.0g
Started | 183 | 182 | 183
Treated | 183 | 182 | 182
Completed | 111 | 119 | 104
Not Completed | 72 | 63 | 79
Not completed — Adverse Event | 20 | 35 | 42
Not completed — Withdrawal by Subject | 11 | 10 | 15
Not completed — Lost to Follow-up | 6 | 3 | 5
Not completed — Lack of Efficacy | 30 | 12 | 13
Not completed — Sponsor Decision | 2 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Xyrem 4.5g | Xyrem 6.0g | Total
Number analyzed (Participants) | 183 | 182 | 183 | 548
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.43) | 47.0 (11.76) | 47.5 (10.61) | 47.0 (11.26)
Age, Customized [Number; unit: participants]
  18 - 39 years | 40 | 57 | 40 | 137
  40 - 49 years | 70 | 47 | 57 | 174
  50 - 64 years | 64 | 69 | 78 | 211
  >=65 years | 9 | 9 | 8 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 166 | 167 | 500
  Male | 16 | 16 | 16 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 6
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 13 | 12 | 33
  White | 167 | 164 | 167 | 498
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 183 | 182 | 183 | 548

OUTCOME MEASURES:

1. Primary Outcome: Pain VAS (Visual Analog Scale) Response. Percentage of Subjects With a Greater Than or Equal to 30% Reduction in Pain VAS From Baseline (BOCF).
Description: Percentage of pain VAS responders. Subjects with a >= 30% reduction in pain VAS from baseline to endpoint (week 14) were considered responders; all other subjects were considered non-responders. Missing data were handled using BOCF (Baseline Observation Carried Forward). The pain VAS ranges from 0 (no pain) to 100 (worst imaginable pain). The pain VAS was collected morning, afternoon and evening. Baseline is the average value recorded for the measure during the week prior to the end-of-baseline visit. Endpoint is the average value recorded for the measure during the week prior to week 14.
Time Frame: Baseline to Week 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Xyrem 4.5g | Xyrem 6.0g
Number analyzed (Participants) | 183 | 182 | 183
Percentage of Participants
  Responder | 27.3 | 46.2 | 39.3
  Non - Responder | 72.7 | 53.8 | 60.7
Statistical Analysis 1: Comparison: Placebo vs Xyrem 4.5g vs Xyrem 6.0g; Overall Comparison; Test type: Superiority or Other; p > 0.001, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Xyrem 4.5g; Pairwise comparison of placebo and Xyrem 4.5g; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Xyrem 6.0g; Pairwise comparison of placebo and Xyrem 6.0g; Test type: Superiority or Other; p = 0.015, Chi-squared

ADVERSE EVENTS:
Arm/Group | Placebo | Xyrem 4.5g | Xyrem 6.0g
Serious Adverse Events (participants affected / at risk) | 1/183 | 0/182 | 2/182
Other Adverse Events (participants affected / at risk) | 105/183 | 149/182 | 145/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=183) | Xyrem 4.5g (N=182) | Xyrem 6.0g (N=182)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess Intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=183) | Xyrem 4.5g (N=182) | Xyrem 6.0g (N=182)
Palpatations (Cardiac disorders) | 0 | 4 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 4
Vision Blurred (Eye disorders) | 0 | 2 | 5
Nausea (Gastrointestinal disorders) | 10 | 26 | 39
Vomiting (Gastrointestinal disorders) | 7 | 8 | 19
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 14
Constipation (Gastrointestinal disorders) | 3 | 4 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 2
Fatigue (General disorders) | 5 | 4 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 7 | 8
Nasopharyngitis (Infections and infestations) | 7 | 8 | 8
Sinusitis (Infections and infestations) | 1 | 12 | 8
Urinary Tract Infection (Infections and infestations) | 2 | 7 | 2
Bronchitis (Infections and infestations) | 2 | 4 | 3
Weight Decreased (Investigations) | 1 | 5 | 5
Blood Pressure Increased (Investigations) | 1 | 3 | 4
Weight Increased (Investigations) | 4 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 5 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 7 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3
Headache (Nervous system disorders) | 20 | 27 | 42
Dizziness (Nervous system disorders) | 5 | 24 | 31
Somnolence (Nervous system disorders) | 9 | 4 | 8
Paraesthesia (Nervous system disorders) | 0 | 7 | 5
Migraine (Nervous system disorders) | 4 | 2 | 2
Sinus Headache (Nervous system disorders) | 2 | 4 | 1
Tremor (Nervous system disorders) | 1 | 1 | 4
Disturbance in Attention (Nervous system disorders) | 0 | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 12 | 10
Insomnia (Psychiatric disorders) | 4 | 3 | 9
Depression (Psychiatric disorders) | 4 | 3 | 5
Nightmare (Psychiatric disorders) | 6 | 2 | 3
Abnormal Dreams (Psychiatric disorders) | 2 | 4 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other